CLINICAL TRIAL: NCT04360265
Title: A Long-term Follow-up Study of Patients With MPS IIIA From Gene Therapy Clinical Trials Involving the Administration of ABO-102 (scAAV9.U1a.hSGSH)
Brief Title: Follow-up Study of AAV-Mediated Gene Transfer (UX111; Previously Known as ABO-102) for MPS Type IIIA
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LTFU-ABO-102; 2019-002979-34 (EudraCT Number); UX111-CL302 (Other: Ultragenyx Pharmaceutical Inc); 2023-510392-66-00 (EU CTIS Number)
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Mucopolysaccharidosis IIIA; MPS IIIA; Sanfilippo Syndrome; Sanfilippo A
Keywords: MPS IIIA; Sanfilippo; Gene Therapy
MeSH Terms: conditions — Mucopolysaccharidosis III | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Other): Participants who have participated in a prior clinical trial involving the administration of UX111 (rebisufligene etisparvovec) and are able to comply with onsite scheduled visits and assessments. Select participants may receive adjuvant IM therapy.
  Interventions: Other: No Investigational Product; Drug: Adjuvant Immunomodulatory (IM) Therapy
- Cohort B (Other): Participants who have participated in a prior clinical trial involving the administration of UX111 (rebisufligene etisparvovec) and who cannot participate in Cohort A. Participants will partake in a reduced number of assessments, performed either onsite or at home via a combination of telehealth and home healthcare visits.
  Interventions: Other: No Investigational Product

INTERVENTIONS:
Other: No Investigational Product — No investigational product will be administered in this follow-up trial.
Drug: Adjuvant Immunomodulatory (IM) Therapy — The Principal Investigator and/or caregiver, in consultation with the medical monitor, will determine whether to initiate adjuvant IM therapy. Not all participants may receive IM therapy.
  Arms: Cohort A

SUMMARY:
The main objective of this study is to evaluate the safety/tolerability and efficacy of UX111 (previously known as ABO-102) in participants with Mucopolysaccharidosis IIIA (MPS IIIA).

DETAILED DESCRIPTION:
This is a multicenter, long-term follow-up study of patients with MPS IIIA who have participated in a prior clinical trial involving the administration of UX111 (NCT02716246 and NCT04088734). No investigational product will be provided. At approved sites adjuvant immunomodulatory (IM) therapy may be administered to selected participants. The Principal Investigator and/or caregiver, in consultation with the medical monitor, will determine whether to initiate adjuvant IM therapy. Not all participants may receive IM therapy.

This study was previously posted by Abeona Therapeutics, Inc and was transferred to Ultragenyx in August 2022.

ELIGIBILITY:
Inclusion Criteria:

* Participants that have participated in a prior clinical trial in which they received UX111
* Parent(s)/legal guardian(s) of participant willing and able to complete the informed consent process and comply with study procedures and visit schedule

Exclusion Criteria:

* Planned or current participation in another clinical trial that may confound the safety or efficacy evaluation of UX111 during this study
* Any other situation or medical condition that precludes the participant from undergoing procedures required in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (SAEs) | Up to Year 5
Bayley Scales of Infant and Toddler Development - Third Edition (BSITD-III) Cognitive Raw Score Over Time | Up to Year 5

SECONDARY OUTCOMES:
Cerebrospinal Fluid (CSF) Heparin Sulfate (HS) (Disaccharide) Exposure | Baseline, Up to Month 36
Percent Change From Baseline in Prior Trial in CSF HS | Baseline, Up to Month 36
BSITD-III Receptive Communication Raw Score Over Time | Up to Year 5
BSITD-III Expressive Communication Raw Score Over Time | Up to Year 5
Annualized Percentage Change from Baseline in Prior Trial in Total Cortical Volume | Baseline, Up to Month 36
Survival | Up to Year 5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (4):
- Nationwide Children's Hospital, Columbus, Ohio, United States
- Women's and Children's Hospital, North Adelaide, South Australia, Australia
- Spain (2):
  - Vall d'Hebron Barcelona Campus, Barcelona
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Ultragenyx Transparency Commitment — https://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/